CLINICAL TRIAL: NCT06625619
Title: On the BRINK: PhotoBiomodulation (PBM) for Mucositis in Patients Undergoing Allogeneic Hematopoietic Stem Cell TRansplant (HSCT) - Implementing the Evidence &Amp; Discovering New Knowledge
Brief Title: On the BRINK: PhotoBiomodulation (PBM) for Mucositis in Patients Undergoing Allogeneic Hematopoietic Stem Cell TRansplant (HSCT) - Implementing the Evidence & Discovering New Knowledge
Status: Active, not recruiting | Type: Observational
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 23673; NCI-2024-01324 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23673 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2024-08-23; First posted 2024-10-03 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Hematopoietic and Lymphatic System Neoplasm; Malignant Solid Neoplasm

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group I (Patients): Patients have their medical records reviewed on study.
  Interventions: Other: Non-Interventional Study
- Group II (Nurses): Nurses complete surveys on study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study

SUMMARY:
This study evaluates mucositis and other oral symptoms in patients undergoing photobiomodulation in patients undergoing hematopoietic stem cell transplantation.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Examine mucositis severity, oral pain, taste changes, and xerostomia in patients undergoing PBM, a new standard of care for oral mucositis.

OUTLINE: This is an observational study. Participants are assigned to 1 of 2 groups.

GROUP I: Patients have their medical records reviewed on study.

GROUP II: Nurses complete surveys on study.

ELIGIBILITY:
Inclusion Criteria:

* PATIENTS:

  * Age: ≥ 18 years
  * Undergoing allogeneic HSCT - cases where PBM was used and cases where PBM was not used

NURSES:

* Nurses who administer PBM

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who are undergoing HSCT and nurses who administer PBM
Sampling Method: Non-Probability Sample
Enrollment: 6 (Estimated)
Dates: Start 2024-10-07 (Actual); Primary Completion 2026-11-24 (Estimated); Study Completion 2026-11-24 (Estimated)

PRIMARY OUTCOMES:
Mucositis according to the World Health Organization (WHO) Scale | Up to 22 days or until discharge, whichever came first
  WHO scale is a combined patient-reported and clinician assessed rating scale that ranges from 0 ( no oral mucositis) to IV (Life threatening mucosistis).
Average oral pain | Up to 22 days or until discharge, whichever came first
  Patient is asked to rate their pain on a 0 - 10 scale with 0 being no pain and 10 being the worst possible pain.
Taste | Up to 22 days or until discharge, whichever came first
  Taste according to the Chemotherapy Induced Taste Alteration Scale (CiTAS) which is an 18-item scale that measures four dimensions of taste: decline in basic taste, discomfort, phantogeusia and parageusia, and general taste alterations. Items are stated on a Likert scale 1 - 5 (where 1 = no difficulty or absence of the disturbance and 5 = maximum difficulty or disturbance.
Xerostomia | Up to 22 days or until discharge, whichever came first
  Xerostomia severity (0-10 scale)

CONTACTS AND LOCATIONS:
Overall Officials: Annette Isozaki, MD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States